ID: UMCC NCT03559049

2018.033

Rucaparib and Pembrolizumab for Maintenance Therapy in Stage IV Non-Squamous Non-Small Cell Lung Cancer

# UNIVERSITY OF MICHIGAN CONSENT TO BE PART OF A RESEARCH STUDY

### 1. KEY INFORMATION ABOUT THE RESEARCHERS AND THIS STUDY

Study title: A Phase I/II Multi-site Study of Rucaparib and Pembrolizumab Maintenance Therapy in Stage IV Non-Squamous Non-Small Cell Lung Cancer after Initial Therapy with Carboplatin, Pemetrexed, and Pembrolizumab

Company or agency sponsoring the study: The University of Michigan along with support from Clovis Oncology and MERCK & Co.

Names, degrees, and affiliations of the principal investigator and study coordinator (if applicable):

### **Principal Investigator:**

Angel Qin, MD Department of Internal Medicine, Hematology/Oncology, University of Michigan

### 1.1 Key Study Information

You may be eligible to take part in a research study. This form contains information that will help you decide whether to join the study. All information in this form is important. Take time to carefully review this information. After you finish, you should talk to the researchers about the study and ask them any questions you have. You may also wish to talk to others such as your friends, family, or other doctors about your possible participation in this study. If you decide to take part in the study, you will be asked to sign this form. Before you do, be sure you understand what the study is about.

### 2. PURPOSE OF THIS STUDY

### 2.1 Study purpose:

A new standard of care for patients with stage IV non-squamous Non-small cell lung cancer (NSCLC) without actionable mutations (DNA change that would be expected to affect a patient's response to treatment) is initial therapy with carboplatin, pemetrexed, and pembrolizumab (also referred to as CPP) followed by maintenance therapy with pembrolizumab and pemetrexed in patients who respond to initial CPP.

Other maintenance therapies are being explored to reduce the risk of regrowth of NSCLC after initial therapy. One such combination, proposed in this study is a combination of pembrolizumab and rucaparib. Rucaparib blocks an enzyme in cells called PARP (poly (ADP-ribose) polymerase); in cancer cells, this leads to increased cell death. Furthermore, a combination of rucaparib and immunotherapy has been shown to be more effective in animal models in reducing cancer growth and leading to increased survival of animals bearing cancers. Recently, rucaparib has been approved in the maintenance setting for ovarian cancer.

In May 2017, pembrolizumab was approved by the Food and Drug Administration (FDA) in combination with pemetrexed and carboplatin for patients with metastatic non-squamous NSCLC who have not received any prior treatment.

Rucaparib, a drug that inhibits PARP enzyme, is approved by the FDA for the treatment of BRCA (breast cancer gene) mutant advanced ovarian cancer who have been treated with two or more previous chemotherapy regimens as well as maintenance therapy in ovarian cancer patients who responded to chemotherapy, regardless of BRCA. It is not FDA approved for the treatment of NSCLC.

To date there are no clinical trials testing the combination of rucaparib and pembrolizumab used as maintenance therapy (a therapy meant to help the primary therapy succeed). Therefore, the purpose of this study is to test the effectiveness (how well the drug combination works), safety, and tolerability of the drug combination of oral rucaparib plus pembrolizumab as maintenance therapy in patients stage IV NSCLC after primary therapy with carboplatin/pemetrexed/pembrolizumab (CPP) therapy.

### 3. INFORMATION ABOUT STUDY PARTICIPANTS (SUBJECTS)

Taking part in this study is completely **voluntary**. You do not have to participate if you don't want to. You may also leave the study at any time. If you leave the study before it is finished, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled.

### 3.1 Who can take part in this study?

Adult men or women who have stage IV non-squamous NSCLC.

There are many other inclusion and exclusion criteria which the doctors will use to determine if you can participate in this study. It is important that you discuss your full medical history and all of your medications with your doctor.

### 3.2 How many people (subjects) are expected to take part in this study?

A total of approximately 55 subjects at several institutions will take part in this study, including approximately 28 from the University of Michigan.

### 4. INFORMATION ABOUT STUDY PARTICIPATION

### 4.1 What will happen to me in this study?

The study team will explain the research study and answer any questions you have about the study. If you want to participate in the study, the study team will request you sign the consent form prior to any activities occurring that pertain to the study. Once your consent is obtained, the study team will look through your medical chart, ask you questions, and begin scheduling tests and procedures to determine if you are eligible for the study. The study team will inform you of the types of tests and procedures required before the study begins.

Many of the procedures that will be performed during the study, including routine blood tests, tumor evaluations (radiology scans), physical examinations, vital signs (blood pressure, heart rate, breathing rate, and temperature) and measurement of height and weight, would normally be done as part of your standard of care regardless of study participation. However, some of these may be done more frequently as a result of your participation in this study. Administration of the study drug combination, tissue/blood collection and analysis are solely for research purposes. Tests and procedures that are done more often than your regular medical care because of your study participation and that are solely for research purposes will be identified below. The study staff will inform you of the types of tests and procedures you have to undergo during the study.

### During the study you must:

- Follow the instructions you are given.
- Come to the study center for your visits with the study doctor.
- Tell the study doctor or study staff about any changes in your health and/or medications you are taking.
- Tell the study doctor or study staff if you want to stop being in the study at any time.

**Before starting the study:** Some exams, tests or procedures will be required to find out if you can be in this study. If you have had some of them recently, they may not need to be repeated. The screening tests and procedures do not have to be completed in one day and you are allowed to take breaks if you have multiple procedures in one day.

The following tests and procedures will be performed during screening and/or at one or more study visits. Refer to the study calendar below for information about which procedures will be performed at certain study visits.

- Vital signs: Including measurement of your height, weight, blood pressure, heart rate, respiratory rate, and temperature.
- Medical history: Including any past treatments, surgeries, infection and autoimmune diseases. You will
  also be asked about medications, and it is important that you tell your doctor about all of the medications
  that you have been taking, including over the counter medicines, vitamins or herbal treatments.
- Physical Exam/Performance Status: Your ability to perform day to day activities and care for yourself.
- Electrocardiogram (ECG): An ECG is a recording of the electrical activity of your heart.
- Urinalysis: A urine sample as an additional method to evaluate your general health.
- Routine blood tests (approximately 2 teaspoons): Will be drawn for tests to check your general health and disease status.
- Pregnancy test (blood approximately 1 teaspoon): Will be drawn if you are a woman able to have children.
- Scans of your cancer: Computed tomography (CT) of the chest and other areas where you have disease.
  - A CT scan uses special x-ray equipment to make detailed pictures of body tissues and organs. For the CT scan, you may be given a "contrast material" (a special dye that makes it easier for doctors to see different tissues in your body). You will be asked to lie still and may be asked to hold your breath for a few seconds. The CT scan is done in the Radiology Department and takes about half an hour.
- Toxicity evaluation: You will be asked about any side effects or illnesses you experience.
- Tumor tissue: Your doctor will check to see if you have enough stored tissue sample of your tumor that
  was collected previously. This is for research purposes.
- Blood for Biomarkers (approximately 1 teaspoon): Will be drawn for testing for biomarkers (testing of substances such as proteins that tell us how the drug is working in your body). This is for research purposes.

### Study Intervention (for Research):

If you qualify to participate in the study based on the results of the screening tests and procedures, you will return to the study doctor's clinic.

For this study a cycle is defined as 21 days. Induction intervention:

Study ID: HUM00147516 IRB: IRBMED Date Approved: 11/11/2022 Expiration Date: 10/27/2023

You will receive pembrolizumab, followed by pemetrexed followed by carboplatin, each given through your vein (IV) every three weeks for a maximum of 4 cycles.

### Maintenance intervention:

If after you receive 4 cycles of the combination of pembrolizumab, carboplatin and pemetrexed, your disease is stable or better you will move to the maintenance portion of the study. On Day 1 of each cycle you will receive pembrolizumab given through your vein or port. You will also take rucaparib every day by mouth on days 1-21 of the cycle. You will continue to take rucaparib and receive pembrolizumab as long as you are tolerating the investigational study treatment and your disease hasn't progressed.

The researchers will ask you to complete a drug diary to track when you have taken your rucaparib. Please bring your drug diary and medication bottles (with extra tablets) with you when you return for each appointment.

### Below are general rules for taking rucaparib:

- Take rucaparib by mouth twice a day as close as possible to 12 hours apart; preferably at the same time
  every day.
- Take with food or without food.
- Swallow whole (do NOT chew, crush or cut the tablet).
- The medication SHOULD NOT be ingested if broken, cracked or otherwise not intact.
- If you miss a dose (i.e. you do not take it within 4 hours of the scheduled time) DO NOT "make it up". Skip the missed dose and start taking rucaparib with the next scheduled dose.
- If you vomit any time after taking a dose DO NOT "make it up".

If you experience side effects, you might have to stop taking all of some of the study drugs and if you recover from your adverse events, you may be able to restart the study drugs.

### Follow-up:

If you stop the study drugs for any reason you will be asked to return for end of treatment visit 30 days after your last dose of study drug.

If you stopped the study drugs for reasons other than disease progression; you will be asked to return to the clinic approximately every 12 weeks to assess your disease status. You will continue to be followed for your disease status until disease progression or you start another anti-cancer intervention.

If your disease progresses information about you will be obtained through your medical records for up to 5 years.

See the table for a summary of the study intervention and procedures.

# Study ID: HUM00147516 IRB: IRBMED Date Approved: 11/11/2022 Expiration Date: 10/27/2023

# Study Procedures Table:

| Follow- | ď | | 2 | | | | | | | 2 | | | | | | × | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Disease | status | Follow-up | | | | | | | | X (every 12 weeks) | | | | | | | | |
| End of | Treatment | Visit | X | X | X | X | X | | X | X | | | | X | X | | | |
| | Cycle 6+ | Day 1 | X | X | X | X | | | | eafter | | × | | | × | | | |
| | Cycle 5 | Day 1 | X | X | X | X | | | | weeks there | | × | | | × | | | |
| Maintenance Phase | Cycle 4 | Day 1 | X | X | X | X | | | | nd every 12 | | × | | × | × | | | |
| Maintena | Cycle 3 | Day 1 | X | X | X | X | | he study | 8 | 2 months at | | × | | | × | | | |
| | Cycle 2 | Day 1 | X | X | X | X | | Every 6 weeks (i.e. every other cycle) throughout the duration of the study | | r the first 1 | | X | | | × | | | |
| | Cycle 1 | Day 1 | X | X | X | X | | ighout the c | 8 | | | | 9 weeks fo | | × | | X | × |
| | Cycle 4 | Day 1 | X | X | X | X | | cycle) throu | 8 | eeks, every | × | | | | × | | | |
| Induction Phase | Cycle 3 | Day 1 | X | X | X | X | | every other | e e | e first 18 w | × | | | | × | | | |
| Induction | Cycle 2 | Day 1 | X | X | X | X | | veeks (i.e. e | 8 | Every 6 weeks for the first 18 weeks, every 9 weeks for the first 12 months and every 12 weeks thereafter | × | | | | × | | | |
| | Cycle 1 | Day 1 | X | X | X | | | Every 6 v | | Every 6 v | × | | | × | | C. | | |
| Screening | | | X | X | X | X | X | X | X | X | | | X | | × | | | |
| Procedures | | | Medical History | Medication Review | Physical Exam/ Vital signs | Routine blood tests | Urinalysis | Pregnancy test | ECG | Scans/Imaging of your | Induction intervention | Maintenance intervention | Tumor Tissue | Research Blood | Toxicity evaluation | Survival follow-up | | |

Consent Subtitle: UMCC 2018.033 Model Consent Version:09Mar2022 UM Consent Version: 27Jul2022

Page 5 of 24

### OPTIONAL Research Samples Stored for Unspecified Future Use:

Besides the information about the main study, the following information is specific to unspecified future use of identifiable data and/or biospecimens. We would also like your permission to keep some of your blood, tumor tissue and medical information collected in the main study, so that we may study it in future research. The future research may be similar to this study or may be completely different.

You can take part in the main study even if you decide not to let us keep your blood, tumor tissue and medical information for future research.

If you give us permission, we will use your blood, tumor tissue and medical information for future research. Even if you give us permission now to keep some of your blood, tissue and medical information, you can change your mind later and ask us to destroy it. Keep in mind, however, that once we have analyzed your blood and tissue, we may not be able to take the information out of our research.

We may share your blood, tumor tissue and medical information with other researchers, so that they can use it in their research. Their research may be similar to this study or may be completely different. Once we have shared your blood, tissue and medical information with other researchers, we will not be able to get it back. Future use of your identifiable data and/or specimens will be conducted in compliance with applicable regulatory requirements.

You will not find out the results of future research on your blood and tumor tissue samples. If you elect to proceed with the optional post-treatment biopsy, the results of the tests run on the tumor tissue samples will be released to your treating doctor. Allowing us to do future research on your blood, tissue and medical information will not benefit you directly.

Research can lead to new discoveries, such as new tests, drugs, or devices. Researchers, their organizations, and other entities, including companies, may potentially benefit from the future research on your blood, tumor tissue and medical information. You will not have rights to these discoveries or any proceeds from them.

You can make your choice about whether to participate in the Optional substudy (storage of research samples for future use) in Section 12 of the consent.

### 4.2 How much of my time will be needed to take part in this study?

The initial screening visit will take approximately 3-5 hours. Each study visit is expected to take approximately 4-6 hours. This is not much longer than what it would take for standard of care.

### 4.3 When will my participation in the study be over?

The maximum time you will be in the study will depend on how your disease responds to the study intervention and how well you tolerate the study intervention. Your participation may end sooner if you decide to no longer participate, your study doctor feels it is in your best interest to stop your study participation, your disease progresses or the study is ended. You can stop participating at any time. However, if you decide to stop participating in the study, we encourage you to talk to the study doctor and your regular physician first.

### 4.4 What will happen with my information and/or biospecimens used in this study?

Your collected information and biospecimens may be shared with Clovis Oncology and Merck & Co.

Your collected information and biospecimens may also be shared with other researchers, both here or around the world, or with companies. Any sharing is subject to contractual obligations with the Sponsor. Additionally:

 With appropriate permissions, your identifiable collected information and biospecimens may also be shared, and/or,

 Without your additional consent, your identifiable collected information and identifiable biospecimens may be stripped of identifiers and used for future research studies or distributed to another researcher for future research studies.

### 5. INFORMATION ABOUT RISKS AND BENEFITS

# 5.1 What risks will I face by taking part in the study? What will the researchers do to protect me against these risks?

The drugs used in the study may cause certain side effects and discomforts. You may have all, some, or none of the known side effects. There is also a risk that other rare or unknown side effects may occur. Your doctors and nurses will check you closely for side effects, and may give you medicines or other treatments to stop or reduce some of these effects. Some side effects may go away soon after the study medication is stopped, but in some cases, side effects may be serious, long lasting, and/or permanent. There is even a chance that a side effect may cause death. If you have any side effects, it is important that you report them to your study doctor or research staff.

These risks will be minimized by monitoring you carefully. We will provide the usual supportive care that would be routinely given to someone with your condition. If you have side effects from the investigational study treatment, we will make appropriate adjustments as defined by the study protocol. You may need to discontinue the investigational study treatment if the side effects are too serious.

The known or expected risks are:

### Side Effects ASSOCIATED WITH PEMETREXED

The following side effects have been described with pemetrexed use when given as a single agent or in combination with other chemotherapy:

- Nausea, vomiting, diarrhea, or constipation
- Low blood cell counts
- Tiredness (also known as lethargy or fatigue)
- Redness or sores in the mouth, throat, lips or esophagus
- Loss of appetite
- Rash or itching

The following table describes side effects reported with pemetrexed.

| | Side Effects with Pemetrexed | |
|---|---|---|
| Common<br>(occurring in 10% or more<br>of patients) | <ul> <li>Your body's ability to fight infections may be affected (Leukopenia: Decrease in white blood cells in the blood, including low levels of neutrophils)</li> <li>Fatigue or shortness of breath (Anemia: decrease in red blood cells in the blood)</li> <li>More likely to bruise or bleed (Thrombocytopenia: low platelet count)</li> </ul> | <ul> <li>Increase in creatinine (marker of kidney function)</li> <li>Fatigue</li> <li>Nausea</li> <li>Vomiting</li> <li>Loss of appetite</li> <li>Constipation</li> <li>Diarrhea</li> <li>Inflammation of the mouth and lips (Stomatitis)</li> <li>Hair loss</li> </ul> |
| Less common<br>(less than 10% of patients) | <ul> <li>Heartburn</li> <li>Taste alteration</li> <li>Numbness, tingling, and burning sensation in hands and feet (Peripheral neuropathy)</li> <li>Dehydration</li> </ul> | <ul> <li>Abnormal liver tests (may suggest liver damage)</li> <li>Infection</li> <li>Painful, red eyes (Conjunctivitis)</li> <li>Rash</li> <li>Itching</li> </ul> |
| Rare<br>(less than 1% of patients) | <ul> <li>Abnormal heart rhythm (Arrhythmia)</li> <li>Allergic reaction</li> <li>Damage to the nerves affecting movement (Motor neuropathy)</li> </ul> | <ul> <li>Kidney failure (Renal failure)</li> <li>Heart attack (Myocardial infarction)</li> <li>Lung disease (Radiation pneumonitis)</li> </ul> |

### Side Effects ASSOCIATED WITH CARBOPLATIN

When receiving carboplatin, you may experience side effects. Side effects when carboplatin is administered alone are described in the table below.

| | Side Effects with Carboplatin | |
|---|---|---|
| Common (occurring in 10% or more of patients) | <ul> <li>Your body's ability to fight infections may be affected (Leukopenia: decrease in white blood cells in the blood, including low levels of neutrophils)</li> <li>Fatigue or shortness of breath (Anemia: decrease in red blood cells in the blood)</li> <li>More likely to bruise or bleed (Thrombocytopenia: low platelet count)</li> </ul> | <ul> <li>Abnormal kidney test (increase blood urea nitrogen and/or creatinine, may suggest kidney damage)</li> <li>Abnormal liver tests (may suggest liver damage)</li> <li>Electrolyte loss (low blood sodium, potassium, calcium, or magnesium)</li> <li>Generalized pain</li> <li>Feeling weak or lack of energy</li> <li>Nausea</li> <li>Vomiting</li> </ul> |
| Less common<br>(less than 10% of patients) | <ul> <li>Numbness, tingling, and burning sensation in hands and feet (Peripheral neuropathy)</li> <li>Sores in mouth (Mucositis)</li> <li>Hair loss</li> <li>Hearing loss</li> <li>Infection</li> </ul> | <ul> <li>Diarrhea</li> <li>Constipation</li> <li>Allergic reaction (symptoms include rash, hives, redness of the skin, itching, breathing difficulty and decreased blood pressure)</li> </ul> |
| Rare<br>(less than 1% of patients) | <ul><li>Heart failure</li><li>Stroke</li><li>Liver failure</li></ul> | <ul> <li>Blood clot</li> <li>Changes in taste</li> <li>Red blood cells that prevent filtering in the kidneys, which can lead to kidney failure (Hemolytic uremic syndrome)</li> </ul> |

### Side Effects ASSOCIATED WITH PEMBROLIZUMAB

Pembrolizumab is a drug that may treat certain cancers by working with your immune system. Pembrolizumab can cause your immune system to attack normal organs and tissues in many areas of the body and can affect the way they work, which can result in side effects. These side effects may be serious (i.e., causing hospitalization or be life-threatening), may result in death, and/or may occur after you stop taking pembrolizumab. These side effects can affect more than one of your normal organs and tissues at the same time.

The following side effects may be caused by pembrolizumab.

<u>VERY COMMON, SOME MAY BE SERIOUS</u> (i.e. causing hospitalization, life-threatening or where noted, may cause death)

Out of 100 people who receive pembrolizumab, 20 or more people may have the following:

- Itching of the skin
- Cough
- Loose or watery stools

<u>COMMON, SOME MAY BE SERIOUS</u> (i.e. causing hospitalization, life-threatening, or where noted, may cause death)

Out of 100 people who receive pembrolizumab, at least 5 but less than 20 people may have the following:

- Joint pain
- Fever
- Back pain
- Rash
- Belly pain
- Loss of skin color
- Not enough thyroid hormone so you may feel tired, gain weight, feel cold, or have infrequent or hard stools (hypothyroidism)
- Low levels of salt in the blood that may cause you to feel tired, feel confused, have a headache, have muscle cramps and/or feel sick to your stomach (hyponatremia)

<u>UNCOMMON, SOME MAY BE SERIOUS</u> (i.e. causing hospitalization, life-threatening, or where noted, may cause death)

Out of 100 people who receive pembrolizumab, at least 1 but less than 5 people may have the following:

- Inflammation of the lungs so you may feel short of breath and cough (pneumonitis)
- Inflammation of the bowels/gut that may cause severe pain in your belly with loose or watery stools, and black, tarry, sticky stools, or stools with blood or mucus (colitis)
- Too much thyroid hormone so you may feel anxious, feel angry, have trouble sleeping, feel weak, tremble, sweat, feel tired, have loose and watery stools (hyperthyroidism)
- Infusion reaction, where you may feel dizzy or faint, feel flushed, get a rash, have a fever, feel short of breath, experience a decrease in your blood pressure at the time of receiving your infusion (IV) or just after, or have pain at the site of infusion
- Inflammation of the skin so you may have peeling of the skin, itchiness, and/or skin redness. The skin
  inflammation (i.e. peeling, itching, and redness) could also be widespread throughout your body. More
  severe skin reactions may involve the inside of your mouth, the surface of your eye and genital areas,
  and/or may cause the top layer of your skin to peel from all over your body which can cause severe
  infection. (Severe skin reactions, including Stevens-Johnson syndrome/or toxic epidermal necrolysis)

RARE, SOME MAY BE SERIOUS (i.e. causing hospitalization, life-threatening, or where noted, may cause death)

Out of 100 people who receive pembrolizumab, less than 1 person may have the following:

- Inflammation of the liver that may make you feel sick to your stomach and vomit, feel like not eating, feel tired, have a mild fever, a pain in the right side of your belly, yellow eyes and skin, and dark urine (hepatitis)
- Inflammation of the pituitary gland (a gland in the head) which may cause you to feel sick to your stomach or have headaches, changes in your behavior, double vision, few to no menstrual cycles, weakness, vomiting and dizziness or fainting (hypophysitis)
- Inflammation of the kidney so you may pass less urine or have cloudy or bloody urine, swelling and low back pain (nephritis)
- Inflammation of the muscles so you may feel weak or pain in the muscles (myositis)
- Inflammation of the pancreas (a gland in your abdomen that controls sugar levels) so you may have severe pain in the top part of your belly that may move to your back, feel sick to your stomach, and have vomiting that gets worse when you eat (pancreatitis)
- Inflammation of the eye so you may have eye redness, blurred vision, sensitivity to light, eye pain, see floaters, or have headaches (uveitis)
- Adrenal glands (glands on top of the kidneys) that may not make enough hormone, which could cause tiredness, weight loss, muscle weakness, feeling faint, having joint, muscle and abdominal aches, nausea, vomiting, loose or watery stools, fever, salt craving, and sometimes darkening of the skin like a suntan (adrenal insufficiency)
- Inflammation of the nerves that may cause pain, weakness, or tingling in your hands and feet, and may spread to your legs, arms and upper body leading to severe muscle weakness and possible temporary paralysis (Guillain-Barre syndrome)
- Type 1 Diabetes, a condition that can cause too much sugar in your blood, feeling thirstier than usual, frequent urination, and weight loss. You are likely to need regular insulin shots
- Inflammation of the middle layer of your heart wall that may cause your heart to have difficulty pumping blood throughout your body, which can cause chest pain, shortness of breath, and swelling of the legs.
   You may experience a fast or irregular heartbeat that may cause you dizziness or fainting (myocarditis)
- Inflammation of the thyroid gland, an organ that makes and stores thyroid hormones. This condition may lead to change in your heart rate, blood pressure, body temperature, and the rate at which food is converted into energy (thyroiditis)
- A condition that may make you feel week and tired and may cause drooping of the eyelids, blurred or double vision, difficulty swallowing, slurred speech, weakness in your arms, and legs or difficulty breathing (myasthenic syndrome/myasthenia gravis including exacerbation)
- The formation of small clusters of immune cells (called granulomas) in parts of your body such as your lymph nodes, eyes, skin or lungs (sarcoidosis)
- Inflammation of the brain with confusion and fever. This may also include: disorientation, memory
  problems, seizures (fits), changes in personality and behavior, difficulty speaking, weakness or loss of
  movement in some parts of your body, and loss of consciousness (encephalitis)
- Inflammation of the spinal cord with pain, numbness, tingling, or weakness in the arms or legs, bladder or bowel problems including needing to urinate more frequently, urinary incontinence, difficulty urinating, and constipation (myelitis)

Additionally, since pembrolizumab was approved in September 2014, the following side effects have been reported by people receiving pembrolizumab. These side effects were voluntarily reported from a group of people of unknown size. It is not possible to estimate the frequency of this side effect:

- Inflammation of the joints which may include joint pain, stiffness and/or swelling (arthritis)
- Severe responses of the immune system that cause the body to attack its own blood cells, spleen, liver, lymph nodes, skin and brain. This may include fever, rash, inflammation of the liver, yellowing of the skin,

- an enlarged liver and spleen, low blood counts, and enlarged lymph nodes. The nervous system may also be affected and cause confusion, seizures, and even coma (hemophagocytic lymphohistiocytosis)
- Changes in eyesight, eye pain, whitish patches on the skin and hearing loss (Vogt-Koyanagi-Harada syndrome)

If you have had an allogeneic stem cell transplant (a procedure in which a person receives blood-forming stem cells from a donor), you may experience graft versus host disease (GvHD), which may include diarrhea, skin rashes, and liver damage, after receiving pembrolizumab. Sometimes this condition can lead to death.

If you have had a solid organ transplant (for example, if you have received a kidney or heart transplant), you may experience rejection of the transplanted organ. Your doctor will monitor you and should tell you what signs and symptoms you should report depending on the type of organ transplant that you have had.

### Side Effects ASSOCIATED WITH RUCAPARIB

Oral rucaparib is an FDA approved drug for patients with ovarian, fallopian and primary peritoneal cancers but considered an experimental drug for lung cancer and therefore may have side effects that cannot be predicted at this time. Rare or unknown side effects could possibly occur, including life-threatening events or death. If you experience certain side effects, your study doctor may decide to stop or lower your dose of study drug until you recover from the side effects.

The following is a list of the most commonly-reported side effects and other notable side effects considered to be possibly due to rucaparib, as reported by physicians about their patients who are taking rucaparib alone:

### Very Common (Occurring in 10% or more of patients)

- Nausea
- Feeling tired
- Changes in kidney and liver function blood tests. These changes will be evaluated by your study team
  along with any other side effects that you are experiencing as well as other test results.
- Changes in your sense of taste
- Low blood counts, (red blood cells, white blood cells, and platelets).
  - A low red blood cell count may make you feel tired or dizzy. If you feel dizzy while taking rucaparib, you should avoid potentially hazardous tasks such as driving or operating machinery.
  - A low white blood cell count puts you at higher risk for bacterial or viral infection. Having a high temperature or fever (a temperature of 100.4°F or 38.0°C) while your white blood cell count is low is a medical emergency and you must proceed to the nearest emergency room as soon as possible.
  - A low platelet count affects the ability of your blood to clot and could lead to bleeding events.
     Symptoms include but are not limited to, easy bruising, prolonged bleeding from cuts, blood in stools or urine, or nose bleeding.
- Stomach-related effects such as, constipation, vomiting, diarrhea, decreased appetite, stomach pain (epigastric pain), and indigestion.
- Increase in cholesterol while taking rucaparib. If your cholesterol increases significantly, your doctor may prescribe a medicine to lower your cholesterol level.
- A low phosphate level in your blood. Usually there are no symptoms but if the levels are critically low, you may notice trouble breathing, confusion, muscle weakness and/or irritability.

- Dizziness
- Difficulty breathing (dyspnea)
- Photosensitivity reaction
  - It is possible that rucaparib may make your skin and eyes more sensitive to sunlight. You should take all of the usual sun protection precautions when going outside. It is advised that you avoid excessive sun exposure, wear protective clothing (including wearing a hat and sunglasses), and use sunscreens regularly (sun protection factor 50 or greater).
- Fever sometimes can occur independent of a low blood count. If you experience an elevation of your temperature, please refer to your study physician for fever management.
- Difficulty sleeping

### Common (Occurring in 1% to less than 10% of patients)

- Rash (also known as dermatitis) which will appear as changes in your skin color (e.g. redness) and texture (e.g. bumps, blisters, peeling). Some rashes may be itchy, painful, or cause no symptoms at all. This can vary in severity from mild to severe. In any case, please inform your study doctor immediately.
- Indigestion
- Itchy skin (also known as pruritus)
- Upper airway infection (like the common cold)
  - You may experience infections involving the nose, pharynx, larynx, and sinuses. Symptoms
    include a blocked (congested) nose, a runny nose, and sneezing. You may also have clear
    discharge (mucus) from the nose. You may feel generally unwell and may also be associated
    with fever. Treatment is usually supportive, but if symptoms persist please inform your
    doctor.

### Uncommon (Occurring in 0.1% up to less than 1% of patients)

Myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML) have been reported in a very small number of patients treated with rucaparib during the safety period (while on treatment with rucaparib and 28 days after last dose). MDS is a pre-cancerous condition where the bone marrow is not as good at producing blood cells (red and/or white blood cells and/or platelets). People with MDS may need transfusions (red blood cells and/or platelets) and/or other treatments. In some cases, MDS can progress to AML, which is a cancer of the bone marrow where more abnormal and immature white blood cells (also called blasts) are made than normal white blood cells. People with AML need treatment with chemotherapy and/or a bone marrow transplant. Patients may develop AML without first being diagnosed with MDS.

Events of MDS and AML have also been reported with PARP inhibitors similar to rucaparib. At this time, it is not known whether rucaparib or other PARP inhibitors cause MDS or AML, or if these developed as a result of previous chemotherapy these patients received. Your Study Doctor will closely monitor your blood cell levels during investigational study treatment. If he/she has any concerns about your blood counts you may be asked to have a biopsy of your bone marrow.

### Allergic Reactions

As with any drug, it is possible that you could have allergic reactions to study drug, such as itching, skin rash, facial swelling, and/or a severe or sudden drop in blood pressure. A sudden drop in blood pressure could lead to shock with loss of consciousness and/or possible seizures, including the possibility of death. If you have any of the above symptoms, seek medical attention right away.

### Risks of CT Scan

The contrast substance injected during the CT scan may cause pain, burning feeling, sweating and rarely a severe allergic reaction that can be serious. If you know you're allergic to iodine you must inform your doctor immediately. The contrast agent used in the CT scan may cause kidney damage, especially if you're diabetic, dehydrated and if you're older. In addition, your thyroid function may be affected. Please inform your doctor if this is the case.

CT imaging uses ionizing radiation, which increases your risk to develop cancer. Everyone is exposed to naturally occurring ionizing radiation every day. The amount of radiation exposure from 1 CT scan is approximately comparable to 1-3 years of natural background radiation. The estimated additional lifetime risk of developing a fatal cancer from a standard CT scan is approximately 1 in 2,000.

### Electrocardiogram (ECG)

An ECG shows the electrical activity of the heart by placing several small adhesive pads that are attached to wires on your chest and limbs (called leads) and connecting them to a machine that reads the signal. There may be minor discomfort, similar to removing a bandage, when the electrodes taped to your chest are removed.

### **Blood tests**

Blood samples will be taken from a vein in your arm during the study. The taking of a blood sample may cause some discomfort and bruising, and there is a potential for infection. Other risks, although rare, include dizziness and fainting.

### Research samples/Loss of Confidentiality

Your samples will be coded, however, there is a risk of loss of confidentiality of your information. If your samples are provided to research collaborators the following information may be made available: your diagnosis and treatments, the time the samples were collected in relation to your study regimen, your disease status, and demographic data (for example gender, race, age, etc.). See section 9 of this document for more information on how the study team will protect your confidentiality and privacy.

### Pregnancy

Taking the study interventions may involve unknown risks to a fetus (unborn baby) if pregnancy were to occur during the study.

If you are a woman of child bearing potential, you must not have sexual intercourse or you must use a reliable form of birth control throughout the study and 180 days after the last dose of study drug. The study doctor will discuss methods of birth control with you if needed. If you choose to use an oral contraception you need to start taking the oral contraception at least 14 days prior to starting the study interventions.

If you are pregnant or become pregnant or are nursing a child during the study, there may be risks to your unborn baby or nursing child. Some drugs cause premature (early) birth or birth defects. Nobody knows what all of these risks are right now.

If you become pregnant or think you may be pregnant during the study, immediately stop using the study drugs and contact the study doctor's office **immediately**. You must not breast-feed an infant during the study. Please also inform the study doctor if you become pregnant up to 180 days after the completion of the study drug. If there is ANY chance that you can get pregnant, you must either agree to not have vaginal intercourse or you must use acceptable birth control (see below).

You must use acceptable birth control for medical reasons all during investigational study treatment (including during temporary breaks from investigational study treatment), and for at least 180 days after investigational study treatment has stopped. You must talk to the doctor before changing any birth control methods you have already agreed to use.

Acceptable methods of contraception are:

Single method (one of the following is acceptable):

- intrauterine device (IUD)
- intrauterine hormone-releasing system (IUS)
- bilateral tubal occlusion
- vasectomy of a female subject's male partner
- contraceptive rod implanted into the skin

Combination method (requires use of two of the following):

- diaphragm with spermicide (cannot be used in conjunction with cervical cap/spermicide)
- cervical cap with spermicide (nulliparous women only)
- contraceptive sponge (nulliparous women only)
- male condom or female condom (cannot be used together)
- hormonal contraceptive: oral contraceptive pill (estrogen/progestin pill or progestin-only pill)
  associated with inhibition of ovulation, contraceptive skin patch, vaginal contraceptive ring, or
  subcutaneous contraceptive injection

Any birth control method can fail. The reports of birth control failing are more frequent for female patients who use only a single form of birth control. Using two forms of birth control at the same time greatly reduces the chances of pregnancy.

### MEN

All men must use an acceptable form of birth control while taking part in the study and for 180 days after investigational study treatment has stopped because the effects on sperm are not known. Acceptable forms of birth control are noted above. Also, men should not donate sperm or semen while taking part in the study and for 180 days after investigational study treatment has stopped because the effects on sperm are not known.

The study doctor must follow up and document the course and the outcome of all pregnancies, even if you withdraw from the study or if the study has finished. If you or your partner become pregnant during the study, the study doctor or his/her staff will ask to contact you or your partner and the pregnancy physician for information about the pregnancy until the child is born and may share this information with the sponsor.

Let your study doctor know of any questions you have about possible side effects. You can ask the study doctor questions about side effects at any time.

As with any research study, there may be additional risks that are unknown or unexpected.

5.2 What happens if I get hurt, become sick, or have other problems as a result of this research?

The researchers have taken steps to minimize the risks of this study. Even so, you may still have problems or side effects, even when the researchers are careful to avoid them. Please tell the researchers listed in Section 10 about any injuries, side effects, or other problems that you have during this study. You should also tell your regular doctors.

### 5.3 If I take part in this study, can I also participate in other studies?

Being in more than one research study at the same time, or even at different times, may increase the risks to you.

It may also affect the results of the studies. You should not take part in more than one study without approval from the researchers involved in each study.

### 5.4 How could I benefit if I take part in this study? How could others benefit?

You may not receive any personal benefits from being in this study. However, information gained in this study may help future patients who are diagnosed with metastatic NSCLC cancer.

# 5.5 Will the researchers tell me if they learn of new information that could change my willingness to stay in this study?

Yes, the researchers will tell you if they learn of important new information that may change your willingness to stay in this study. If new information is provided to you after you have joined the study, it is possible that you may be asked to sign a new consent form that includes the new information.

### 6. OTHER OPTIONS

### 6.1 If I decide not to take part in this study, what other options do I have?

You do not have to be in this study to get treatment for your cancer. Other possible options include:

- Treatment with standard of care drugs such as platinum-based chemotherapy alone or targeted oral pills such as afatinib, erlotinib, gefitinib, osimertinib crizotinib, ceritinib, alectinib, brigatinib, trametinib and dabrafenib.
- You could participate in other research trials
- You could receive palliative radiation
- You could choose not to receive any treatment

You should talk to your study doctor and your regular physician about each of your options and their risks and benefits before you decide if you want to take part in this study.

### 7. ENDING THE STUDY

### 7.1 If I want to stop participating in the study, what should I do?

You are free to leave the study at any time. If you leave the study before it is finished, there will be no penalty to you. You will not lose any benefits to which you may otherwise be entitled. If you choose to tell the researchers why you are leaving the study, your reasons for leaving may be kept as part of the study record. If you decide to leave the study before it is finished, please tell one of the persons listed in Section 10 "Contact Information" (below).

### 7.2 Could there be any harm to me if I decide to leave the study before it is finished?

If you decide to leave the study early, please notify someone on the study team. They will instruct you on how to stop the study safely and you will be advised whether any additional test may need to be done for your safety.

### 7.3 Could the researchers take me out of the study even if I want to continue to participate?

Yes. There are many reasons why the researchers may need to end your participation in the study. Some examples are:

- √ The researcher believes that it is not in your best interest to stay in the study.
- ✓ You become ineligible to participate.
- ✓ Your condition changes and you need treatment that is not allowed while you are taking part in the study.
- ✓ You do not follow instructions from the researchers.
- √ The study is suspended or canceled.

### 8. FINANCIAL INFORMATION

**8.1** Who will pay for the costs of the study? Will I or my health plan be billed for any costs of the study? The study will pay for research-related items or services that are provided only because you are in the study. If you are not sure what these are, see Section 4.1 above or ask the researchers for a list. If you get a bill you think is wrong, call the researchers' number listed in section 10.1.

Rucaparib will be provided by Clovis Oncology free of charge.

Pembrolizumab will be provided by Merck free of charge.

You or your health plan will pay for all the things you would have paid for even if you were not in the study, like:

- Pemetrexed and carboplatin
- Health care given during the study as part of your regular care
- Items or services needed to give you study drugs or devices
- Monitoring for side effects or other problems
- Deductibles or co-pays for these items or services

If you do not have a health plan, or if you think your health plan may not cover these costs during the study, please talk to the researchers listed in Section 10 below or call your health plan's medical reviewer.

"Some health plans will not cover the cost of standard treatments when they are combined with investigational treatments. It is important that you work with the study team to confirm your health plan will cover the costs of carboplatin/pemetrexed/pembrolizumab if you take part in this study."

The study team has given you instructions about this research study. It is important that you follow these instructions carefully. If you get sick, have a medical complication, or are injured as a result of your being in the study, call Dr. Qin, at 734-936-4000 (24-hour Hospital Paging Operator). The doctor will either treat you or send you to another doctor for treatment.

You will get free hospitalization or emergency room care at the UMHS for any immediate complication, injury, or illness caused by the study drug, device, or procedure. The UMHS and the study doctor are responsible for determining whether your condition was the result of your participation in the study.

The UMHS will pay for your hospitalization or emergency room visit only if the need for treatment has been caused by the study drug, device or procedure. This means that you or your health plan must pay for any treatment that is part of your usual medical care or that is related to a medical condition you had before participating in the study.

By signing this form, you do not give up your right to seek payment if you are harmed as a result of being in this study.

## 8.2 Will I be paid or given anything for taking part in this study?

You will not be paid to take part in this study.

### 8.3 Who could profit or financially benefit from the study results?

Information obtained from this study may help the supporters Merck and Clovis Oncology and/or the University of Michigan learn more about the causes, risks, treatments, or how to prevent this and other health problems.

Merck, Clovis Oncology the University of Michigan, or physicians at the university could profit financially from this information.

Research can lead to new discoveries, such as new tests, drugs, or devices. Researchers, their organizations, and other entities, including companies, may potentially benefit from the use of the data or discoveries. You will not have rights to these discoveries or any proceeds from them.

# 9. CONFIDENTIALITY OF SUBJECT RECORDS AND AUTHORIZATION TO RELEASE YOUR PROTECTED HEALTH INFORMATION

The information below describes how your privacy and the confidentiality of your research records will be protected in this study.

### 9.1 How will the researchers protect my privacy?

The University of Michigan has rules to protect information about you. Federal and state laws also protect your privacy. Upon enrolling in this study, you will be assigned a unique identification number. All records and research blood samples related to the study will use this identification number instead of your name or other personally identifying information whenever possible. We will take measures to protect the privacy and security of all your personal information, but we cannot guarantee complete confidentiality of study data.

Medical information created by this research study may become part of your hospital medical record and may be forwarded to your primary doctor. Information that does not become part of your medical record will be stored in your study file.

You have the right to request access to your protected health information that is used or shared during this research and that is related to your study treatment for your study treatment, but you may access this information only after the study is completed. To request this information, please contact the researchers listed in Section 10 "Contact Information" (below).

### **Genetic Risks:**

The federal Genetic Information Nondiscrimination Act (GINA) generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. Under this law:

- Health insurance companies and group health plans may not request your genetic information that we obtain from this research
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums
- Employers with 15 or more employees may not use your genetic information that we obtain from this
  research when making a decision to hire, promote, or fire you or when setting the terms of your
  employment

GINA does not apply to the following groups; however, these groups have policies in place that provide similar protections against discrimination:

- Members of the US Military receiving care through Tricare
- Veterans receiving care through the Veteran's Administration (VA)
- The Indian Health Service
- Federal employees receiving care through the Federal Employees Health Benefits Plans

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

9.2 What information about me could be seen by the researchers or by other people? Why? Who might see it? Signing this form gives the researchers your permission to obtain, use, and share information about you for this study, and is required in order for you to take part in the study. Information about you may be obtained from any hospital, doctor, and other health care provider involved in your care, including:

- Hospital/doctor's office records, including test results (X-rays, blood tests, urine tests, etc.)
- Mental health care records (except psychotherapy notes not kept with your medical records)
- Alcohol/substance abuse treatment records
- HIV/AIDS status
- Sexually transmitted disease or other communicable disease status
- Health plan/health insurance records
- All records relating to your condition, the treatment you have received, and your response to the treatment
- Billing information
- Demographic information
- Personal information

There are many reasons why information about you may be used or seen by the researchers or others during or after this study. Examples include:

- The researchers may need the information to make sure you can take part in the study.
- The researchers may need the information to check your test results or look for side effects.
- University of Michigan, Food and Drug Administration (FDA), and/or other government officials, auditors, and/or the IRB may need the information to make sure that the study is done in a safe and proper manner.
- Merck, Clovis Oncology or safety monitors or committees, may need the information to:
  - Make sure the study is done safely and properly
  - Learn more about side effects
  - Analyze the results of the study
- Insurance companies or other organizations may need the information in order to pay your medical bills or other costs of your participation in the study.
- The researchers may need to use the information to create a databank of information about your condition or its treatment.
- Information about your study participation may be included in your regular University of Michigan medical record.
- Federal or State law may require the study team to give information to government agencies. For example, to prevent harm to you or others, or for public health reasons.

The results of this study could be published in an article, but would not include any information that would let others know who you are.

### 9.3 What happens to information about me after the study is over or if I cancel my permission?

As a rule, the researchers will not continue to use or disclose information about you, but will keep it secure until it is destroyed. Sometimes, it may be necessary for information about you to continue to be used or disclosed, even after you have canceled your permission or the study is over.

Examples of reasons for this include:

- To avoid losing study results that have already included your information
- To provide limited information for research, education, or other activities (This information would not include your name, social security number, or anything else that could let others know who you are.)
- To help the University of Michigan and government officials make sure that the study was conducted properly

As long as your information is kept within the University of Michigan Health System, it is protected by the Health System's privacy policies. For more information about these policies, ask for a copy of the University of Michigan "Notice of Privacy Practices". This information is also available on the web at

http://www.uofmhealth.org/patient+and+visitor+guide/hipaa. Note that once your information has been shared with others as described under Question 9.2, it may no longer be protected by the privacy regulations of the federal Health Insurance Portability and Accountability Act of 1996 (HIPAA).

### 9.4 When does my permission expire?

Your permission expires at the end of the study, unless you cancel it sooner. You may cancel your permission at any time by writing to the researchers listed in Section 10 "Contact Information" (below).

### 10. CONTACT INFORMATION

### 10.1 Who can I contact about this study?

Please contact the researchers listed below to:

- Obtain more information about the study
- · Ask a question about the study procedures or treatments
- Talk about study-related costs to you or your health plan
- Report an illness, injury, or other problem (you may also need to tell your regular doctors)
- Leave the study before it is finished
- Express a concern about the study



You may also express a concern about a study by contacting the Institutional Review Board listed below.

University of Michigan Medical School Institutional Review Board (IRBMED)

2800 Plymouth Road

Building 520, Room 3214

Ann Arbor, MI 48109-2800



If you are concerned about a possible violation of your privacy or concerned about a study you may contact the University of Michigan Health System Compliance Help Line at 1-866-990-0111.

When you call or write about a concern, please provide as much information as possible, including the name of the researcher, the IRBMED number (at the top of this form), and details about the problem. This will help University

Study ID: HUM00147516 IRB: IRBMED Date Approved: 11/11/2022 Expiration Date: 10/27/2023

officials to look into your concern. When reporting a concern, you do not have to give your name unless you want to.

### 11. RECORD OF INFORMATION PROVIDED

### 11.1 What documents will be given to me?

You will receive a copy of the signed and dated informed consent

Your signature in the next section means that you have received copies of all of the following documents:

- This "Consent to be Part of a Research Study" document.
- Other (specify):

| 12. SIGNATURES |
|---|
| Consent/Assent to Participate in the Research Study |
| I understand the information printed on this form. I have discussed this study, its risks and potential benefits, and my other choices with My questions so far have been answered. I understand that if I have more questions or concerns about the study or my participation as a research subject, I may contact one of the people listed in Section 10 (above). I understand that I will receive a copy of this form at the time I sign it and later upon request. I understand that if my ability to consent or assent for myself changes, I may be asked to re-consent prior to my continued participation in this study. |
| Print Legal Name: |
| Signature: |
| Date of Signature (mm/dd/yy): |
| Consent/Assent to Collect and Store OPTIONAL Research Samples for Unspecified Future Use This project involves the option to allow the study team to keep your identifiable specimens/data for use in future research. I understand that it is my choice whether or not to take part in this optional research. I understand that if my ability to consent or assent for myself changes, I or my legal representative may be asked to re-consent prior to my continued participation in this study. |
| Yes, I agree to let the study team keep and store my blood and tissue samples for future research. |
| No, I do not agree to let the study team keep and store my blood and tissue samples for future research. |
| Print Legal Name: |
| Signature: |
| Date of Signature (mm/dd/yy): |

| Principal Investigator or Designee |
|---|
| I have provided this participant and/or his/her legally authorized representative(s) with information about this study that I believe to be accurate and complete. The participant indicated that he or she understands the nature of the study, including risks and benefits of participating. |
| Legal Name: |
| Title: |
| Signature: |
| Date of Signature (mm/dd/yy): |

| U of M Study # | <u> </u> |
|----------------|----------|
|----------------|----------|

Namo

# PERSONAL CENSUS FORM

Data

| IVG | | | |
|---|---|---|---|
| Ce | ne National Cancer Institute requires that The<br>enter report race and ethnicity information ab<br>sure that all populations are offered the oppo | out pe | ople who participate in clinical research to |
| | Check here if you do not wish to provide sor | ne or a | Ill of the information below. |
| 1. | What race do you consider yourself to be? (Please select one or more) | 0000 | American Indian/Alaska Native <sup>a</sup> Asian <sup>b</sup> Black or African American <sup>c</sup> Native Hawaiian or Other Pacific Islander <sup>d</sup> White <sup>e</sup> More than one race <sup>f</sup> |
| 2. | Do you consider yourself to be Hispanic <sup>9</sup> ? | □ Ye | s □ No |

<sup>&</sup>lt;sup>a</sup> American Indian or Alaska Native- A person having origins in any of the original peoples of North, Central, or South America, and who maintains tribal affiliation or community attachment.

<sup>&</sup>lt;sup>b</sup> Asian- A person having origins in any of the original peoples of the Far East, Southeast Asia, or the Indian subcontinent, including, for example, Cambodia, China, India, Japan, Korea, Malaysia, Pakistan, the Philippine Islands, Thailand and Vietnam.

<sup>&</sup>lt;sup>c</sup> Black or African American- A person having origins in any of the black racial groups of Africa. (Terms such as "Haitian" or "Negro" are sometimes used in addition to "Black" or "African American.")

<sup>&</sup>lt;sup>d</sup> Native Hawaiian or Other Pacific Islander- A person having origins in any of the original peoples of Hawaii, Guam, Samoa, or other Pacific Islands.

<sup>&</sup>lt;sup>e</sup> White- A person having origins in any of the original peoples of Europe, the Middle East, or North Africa.

f More than one race- (It is preferred that this be selected in addition to the selection of the specific races listed above, but this may also be solely selected.)

<sup>&</sup>lt;sup>g</sup> Hispanic or Latino- A person of Mexican, Puerto Rican, Cuban, Central or South American, or other Spanish culture or origin, regardless of race. The term "Spanish origin" is sometimes used in addition to "Hispanic" or "Latino."